CLINICAL TRIAL: NCT06210425
Title: Is Re-examination of Urine Culture Necessary for Patients With Preoperative Positive Results in Predicting Infectious Complications Related to Mini-Percutaneous Nephrolithotomy?
Brief Title: Is it Necessary for Patients With a Positive Urine Culture to Achieve a Negative Result After Antimicrobial Treatment Before Undergoing Percutaneous Nephrolithotomy?
Status: Completed | Type: Observational
Sponsor: Junhao Zheng (Other)
Responsible Party: Sponsor-Investigator, Junhao Zheng, Resident, The First Affiliated Hospital of Guangzhou Medical University
Organization: The First Affiliated Hospital of Guangzhou Medical University (Other)
Other Study IDs: 12440100455344205E
Record Dates: First submitted 2024-01-06; First posted 2024-01-18 (Actual); Last update posted 2025-11-21 (Actual); Status verified 2024-01

CONDITIONS: Kidney Calculi; Urinary Tract Infections; Sepsis
Keywords: Percutaneous nephrolithotomy; Urine culture; Antibiotics; Infectious complication; Sepsis
MeSH Terms: conditions — Kidney Calculi; Urinary Tract Infections; Sepsis

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Urine culture
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- Preoperative urine culture positive group: Preoperative urine culture was positive
- Preoperative urine culture negative group: preoperative urine culture was negative

SUMMARY:
Objective: The current European Association of Urology (EAU) guidelines do not provide clear recommendations on whether patients with a positive urine culture(UC) should wait until the culture turns negative following antimicrobial treatment before undergoing percutaneous nephrolithotomy (PCNL). This study evaluates the necessity of achieving a negative UC after treatment with sensitive antibiotics before performing PCNL.

Methods: A prospective, continuous study was carried out involving patients with a positive UC who underwent percutaneous nephrolithotomy (PCNL) at the Department of Urology, The First Affiliated Hospital of Guangzhou Medical University, between March 2021 and April 2024. Patients received treatment with sensitive antibiotics for 5 to 7 days based on the drug susceptibility results of their initial UC upon admission. Follow-up UCs were performed on the third day after starting antibiotic treatment and again immediately before the surgery. An analysis was conducted to examine the relationship between UC results at the two specified time points and the occurrence of infectious complications following PCNL.

DETAILED DESCRIPTION:
For large renal stones, percutaneous nephrolithotomy (PCNL) is the recommended standard surgical approach, especially in cases involving infectious renal stones. Postoperative infections have become the most common complication associated with PCNL, often necessitating additional antimicrobial treatment and prolonged hospitalization. Therefore, it is critically important to identify the risk factors linked to infections after PCNL. Preoperative UC directs antibiotic treatment and mitigates infectious complications post-PCNL. Even with negative preoperative UCs and suitable antibiotic treatment, SIRS or sepsis may still develop post-PCNL. Several studies have indicated that a preoperative UC obtained before antibiotic administration is not a reliable predictor of postoperative infectious complications. Nonetheless, there has been limited research on the relationship between repeat UCs after antibiotic treatment and post-PCNL infectious complications. This research assesses the necessity of achieving a negative UC after treatment with sensitive antibiotics before undergoing PCNL.

ELIGIBILITY:
Inclusion Criteria:

1. Age ≥ 18 years.
2. Renal stone diameter ≥ 2 cm, complex renal stones, or failed ESWL treatment.
3. Consent to undergo PCNL with a positive midstream urine culture preoperatively.
4. ASA score of I or II.

Exclusion Criteria:

1. Coexisting renal tumor.
2. Use of antibiotics within the past two weeks.
3. Renal dysfunction (serum creatinine >451 μmol/L).
4. Unresolved hemorrhage or coagulation abnormalities.
5. Patients who have undergone percutaneous renal fistula or have a ureteral stent in place on the affected side.
6. Simultaneous bilateral renal stone surgery.
7. Severe underlying diseases, such as respiratory or circulatory insufficiency, that cannot tolerate anesthesia or surgery.
8. Pregnant or lactating women.

Ages: 18 Years to 80 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Patients received treatment with sensitive antibiotics for 5 to 7 days based on the drug susceptibility results of their initial UC upon admission. Follow-up UCs were performed on the third day after starting antibiotic treatment and again immediately before the surgery. An analysis was conducted to examine the relationship between UC results at the two specified time points and the occurrence of infectious complications following PCNL.
Sampling Method: Non-Probability Sample
Enrollment: 147 (Actual)
Dates: Start 2021-03-01 (Actual); Primary Completion 2024-10-30 (Actual); Study Completion 2024-11-10 (Actual)

PRIMARY OUTCOMES:
SIRS | Within 7 days postoperatively
  The presence of at least two of the following four criteria defines SIRS following PCNL: heart rate greater than 90/min, white blood cell count ≥12 × 10^9/L or ≤4 × 10^9/L, body temperature above 38°C or under 36°C, and respiratory rate greater than 20/min.
Urosepsis | Within 7 days postoperatively
  ①Confirmed urinary tract infection; ②SOFA (Sequential Organ Failure Assessment) score ≥2 points. A diagnosis of urosepsis can be made if both of the above conditions are met.

CONTACTS AND LOCATIONS:
Locations (1):
- The First Affiliated Hospital of Guangzhou Medical University, Guangzhou, GuangGong, China